CLINICAL TRIAL: NCT04568213
Title: Effect of Hypochlorous Acid Disinfection on Ocular Flora Prior to Cataract Surgery
Brief Title: Hypochlorous Acid Disinfection Prior to Cataract Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Loma Linda University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 5200306
Record Dates: First submitted 2020-09-24; First posted 2020-09-29 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Cataract; Endophthalmitis
Keywords: Ocular/Eyelid Flora
MeSH Terms: conditions — Cataract; Endophthalmitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Hypochlorous Gel Application (Experimental)
  Interventions: Drug: Hypochlorous Acid Gel 0.02%

INTERVENTIONS:
Drug: Hypochlorous Acid Gel 0.02% — 0.02% Hypochlorous Acid Gel (OCusoft Hypochlor GEL) will be sprayed onto the closed eyelid of the surgical eye while covering the fellow eye with palm of the hand, left for 60 seconds, then wiped off with a clean gauze, tissue, or cotton ball.

SUMMARY:
Antibiotics are commonly utilized to reduce the bacterial population of the eye prior to surgery with the assumption that this reduces the risk of endophthalmitis, although it is not clear if this actually occurs. This study will investigate the use of Hypochlorous Acid, a commercially available over the counter (OTC) medication to see if this will reduce the bacterial population prior the cataract surgery.

ELIGIBILITY:
Inclusion Criteria:

- Patients undergoing cataract surgery.

Exclusion Criteria:

* Age <18 years old
* Vulnerable subjects
* Non-English Speakers

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2020-10-29 (Actual); Primary Completion 2022-12-09 (Actual); Study Completion 2022-12-09 (Actual)

PRIMARY OUTCOMES:
Reduction in bacterial flora in eyelashes of treatment eye compared to fellow eye | On day of surgery prior to surgical prep
  Swab will be used to obtain samples from the eyelashes bilaterally and cultured
Reduction in bacterial flora in conjunctiva of treatment eye compared to fellow | On day of surgery prior to surgical prep
  Swab will be used to obtain samples from the conjunctiva bilaterally and cultured

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey J Ing, MD, Principal Investigator — Loma Linda University Department of Ophthalmology
Locations (1):
- Loma Linda University Health, Loma Linda, California, United States

IPD SHARING:
Plan to Share IPD: No